CLINICAL TRIAL: NCT03734094
Title: Comparative Study Between Custom-made Ceramic Barrier and Titanium Mesh for Augmentation of Atrophic Posterior Mandible
Brief Title: Custom-made Ceramic Barrier vs Titanium Mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed El Saharty, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 737
Record Dates: First submitted 2018-11-01; First posted 2018-11-07 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceramic Barrier (Experimental): The use of a ceramic barrier to induce bone formation during GBR
  Interventions: Device: Titanium Mesh
- Titanium mesh (Active Comparator): The use of a titanium mesh to induce bone formation during GBR
  Interventions: Device: Ceramic barrier

INTERVENTIONS:
Device: Ceramic barrier — The use of a ceramic barrier to induce bone formation during GBR
  Arms: Titanium mesh
Device: Titanium Mesh — The use of a titanium mesh to induce bone formation during GBR
  Arms: Ceramic Barrier

SUMMARY:
It is a comparative study between custom-made ceramic barrier and titanium mesh for augmentation of atrophic posterior mandible.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrophic posterior mandible
* Both sexes
* No intraoral soft and hard tissue pathology
* No systemic condition that contraindicate implant placement

Exclusion Criteria:

* Untreated gingivitis
* Periodontitis
* Insufficient oral hygiene
* Previous radiation therapy
* Head and neck neoplasia
* Systemic disorders
* Heavy smokers
* Bone pathology
* Psychiatric problems
* Emotional instability
* Unrealistic aesthetic demands

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Bone height | 6 months
  CBCT & Three dimensional planning software to measure the height of bone gained in millimeters.
Bone width | 6 months
  CBCT & Three dimensional planning software to measure the width of bone gained in millimeters.

SECONDARY OUTCOMES:
Histomorphometric - bone area percent | 6 months
  Histomorphometric analysis of bone area percent

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes